CLINICAL TRIAL: NCT06010017
Title: Peer Support Intervention for Patients Undergoing Hematopoietic Stem Cell Transplantation (STEPP): Feasibility and Preliminary Efficacy Trial
Brief Title: Peer Support Intervention for Patients Undergoing Hematopoietic Stem Cell Transplantation
Acronym: STEPP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Hermioni L.Amonoo, MD, MPP, MPH, Director, Well-Being and Cancer Research Program, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 23-132
Record Dates: First submitted 2023-08-21; First posted 2023-08-24 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Hematopoietic Neoplasms; Hematopoietic Malignancy
Keywords: Hematopoietic Neoplasms; Hematopoietic Malignancy; HSCT; Hematopoietic Stem Cell Transplantation
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- STEPP (Experimental): Participants will be randomized in 1:1 fashion, stratified by transplant type (autologous vs. allogeneic), and will complete study procedures as follows:
  * Baseline self-reported assessment (in-person or remotely).
  * Virtual, STEPP intervention sessions 1x weekly for five weeks with peer mentor.
  * HSCT and hospitalization per standard of care.
  * Day +30 (+/- 10 days) and Day +60 (+/- 10 days) self-reported assessments.
  * Optional exit interview with study staff (40 participants).
  Interventions: Behavioral: STEPP Intervention
- Usual Care (No Intervention): Participants will be randomized in 1:1 fashion, stratified by transplant type (autologous vs. allogeneic), and will complete study procedures as follows:
  * Baseline self-reported assessment.
  * HSCT and hospitalization per standard of care.
  * Day +30 (+/- 10 days) and Day +60 (+/- 10 days) self-reported assessments.

INTERVENTIONS:
Behavioral: STEPP Intervention — Peer support intervention comprised of five learning modules on psychoeducation and supportive psychotherapy strategies, via virtual platform. If participants do not have a smart device, one will be provided by the study team.
  Arms: STEPP

SUMMARY:
The main purpose of this study is to determine if a novel peer support intervention (STEPP) is feasible among patients undergoing hematopoietic stem cell transplantation (HSCT).

The name of the intervention used in this research study is STEPP, a peer support intervention comprised of five learning modules on psychoeducation and supportive psychotherapy strategies, tailored to the unique needs of patients undergoing HSCT.

DETAILED DESCRIPTION:
The goal of this project is to refine a peer support intervention (STEPP) for patients undergoing hematopoietic stem cell transplantation (HSCT) and to conduct a randomized clinical trial to test its feasibility and preliminary efficacy for improving quality of life (QOL) and reducing psychological distress.

Participants will be randomized into one of two study groups: Peer Support Intervention (STEPP) vs. Usual Care. Randomization means a participant is placed into a group by chance. Participants will have an equal chance of being placed in either group.

Study procedures include screening for eligibility and questionnaires.

Participation in this study is expected to last about 10 weeks.

It is expected that about 80 people will participate in this randomized clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age > 18 years) with a hematologic malignancy undergoing autologous or allogeneic HSCT.
* Ability to comprehend, read, and respond to questions in English as STEPP is only available in English.

Exclusion Criteria:

* Patients undergoing HSCT for benign hematologic conditions.
* Patients undergoing outpatient HSCT.
* Patients with acute or unstable psychiatric or cognitive conditions which the treating clinicians believes prohibits informed consent or compliance with study procedures.
* Patients undergoing HSCT for the second time.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2024-02-20 (Actual); Primary Completion 2025-03-03 (Actual); Study Completion 2025-03-21 (Actual)

PRIMARY OUTCOMES:
Feasibility of STEPP | Up to 10 weeks
  The proposed STEPP intervention will be deemed feasible if at least 60% of eligible patients are enrolled in the study, and of those enrolled and randomized to the intervention, at least 60% complete at least 3/5 of the intervention sessions.

SECONDARY OUTCOMES:
Acceptability of STEPP | Up to Day +60 (+/- 10 days)
  The 7-item Client Satisfaction Questionnaire (CSQ) will assess patient satisfaction with the STEPP intervention. Each question is scored from 0-4 to result in a total of 0-28. Higher scores indicate increased acceptability of the intervention.
Anxiety Symptoms based on the Hospital Anxiety and Depression Scale-Anxiety Subscale (HADS-A) | Up to Day +60 (+/- 10 days)
  Compare anxiety symptoms using the Hospital Anxiety and Depression Scale-Anxiety Subscale (HADS-A) between the two groups. The HADS-A is comprised of 7 items that quantify the degree to which participants experience mood symptoms, with each item's score ranging from 0 to 3. Scores range from 0 to 21, with a cutoff of 8 or greater denoting clinically significant anxiety.
Quality of Life based on the Functional Assessment of Cancer Therapy-Bone Marrow Transplant (FACT-BMT) | Up to Day +60 (+/- 10 days)
  Compare quality of life (QOL) using the 45-item Functional Assessment of Cancer Therapy-Bone Marrow Transplant (FACT-BMT) between the two groups.
  The FACT-BMT consists of five subscales assessing well-being across the following domains: physical, functional, emotional, social, and bone marrow transplant symptoms. Each question is scored from 0 ("Not at all") to 4 ("Very Much"). The FACT-BMT ranges from 0 to 148, with higher scores indicating better quality of life.
Depression Symptoms based on the Hospital Anxiety and Depression Scale-Depression Subscale (HADS-D) | Up to Day +60 (+/- 10 days)
  Compare depression symptoms using the Hospital Anxiety and Depression Scale-Depression Subscale (HADS-D) between the two groups. The HADS-D is comprised of 7 items that quantify the degree to which participants experience mood symptoms, with each item's score ranging from 0 to 3. Scores range from 0 to 21, with a cutoff of 8 or greater denoting clinically significant depression.
Post-Traumatic Stress Symptoms based on the Post-traumatic Stress Checklist-Civilian Version (PCL-C) | Up to Day +60 (+/- 10 days)
  Compare post-traumatic stress disorder symptoms using the 17-item Post-traumatic Stress Checklist-Civilian Version (PCL-C) between the two groups.
  The PCL-C evaluates symptoms of post-traumatic stress disorder according to the criteria of the Diagnostic and Statistical Manual of Mental Disorders-IV. Each item is scored from 1 to 5 for a total score ranging from 17 to 85. A higher score indicates greater severity of post-traumatic stress disorder symptoms.
Social Support based on the Social Support Effectiveness Questionnaire (SSEQ) | Up to Day +60 (+/- 10 days)
  Compare social support using the 26-item Social Support Effectiveness Questionnaire (SSEQ) between the two groups.
  The SSEQ is a validated instrument used in the oncological population to assess patients' perception of social support. The total score ranges from 0 to 80, with higher scores indicating more effective support.

OTHER OUTCOMES:
Self-Efficacy based on the Cancer Self-Efficacy Scale-transplant (CASE-t) | Up to Day +60 (+/- 10 days)
  Compare self-efficacy using the Cancer Self-Efficacy Scale-transplant (CASE-t) between the two groups.
  The CASE-t assesses patients' confidence in managing the impact of their illness. Scores range from 0 to 170, with higher scores indicating greater self-efficacy.
Gratitude based on the Gratitude Questionnaire | Up to Day +60 (+/- 10 days)
  Compare gratitude using the 6-item Gratitude Questionnaire between the two groups.
  The Gratitude Questionnaire ranges from 6 to 42, with higher scores indicating a stronger propensity for experiencing gratitude in daily life.
Positive Affect based on the Positive and Negative Affect Schedule Positive Affect Subscale | Up to Day +60 (+/- 10 days)
  Compare positive affect using the 10-item Positive Affect Subscale from the Positive and Negative Affect Schedule (PANAS) between the two groups.
  The Positive Affect Subscale ranges from 10 to 50, with higher scores indicating higher levels of positive affect.
Flourishing based on the Flourishing Scale | Up to Day +60 (+/- 10 days)
  Compare flourishing using the 8-item Flourishing Scale between the two groups.
  The Flourishing Scale ranges from 8 to 56, with higher scores indicating having more psychological resources and strengths.

CONTACTS AND LOCATIONS:
Overall Officials: Hermioni Amonoo, MD, MPP, MPH, Principal Investigator — Brigham and Women's Hospital
Locations (2):
- United States (2):
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber/Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to Sponsor, Investigator, or designee. The protocol and statistical analysis plan will be made available on ClinicalTrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the study investigator at hermioni_amonoo@dfci.harvard.edu

REFERENCES:
- [Derived] Keane EP, Guo M, Gudenkauf LM, Boardman AC, Song MT, Wolfe ED, Larizza IS, Mate-Kole MN, Healy BC, Huffman JC, El-Jawahri A, Amonoo HL. A peer support intervention in patients with hematologic malignancies undergoing hematopoietic stem cell transplantation (HSCT): The STEPP randomized pilot trial design and methods. Contemp Clin Trials. 2025 Jan;148:107746. doi: 10.1016/j.cct.2024.107746. Epub 2024 Nov 19. PMID 39566722